CLINICAL TRIAL: NCT02644148
Title: The Effect of Uncut Roux-en-Y Gastrojejunostomy on Quality of Life After Laparoscopic Distal Gastrectomy for Early Gastric Cancer Patients
Brief Title: Uncut Roux-en-Y Gastrojejunostomy for Early Gastric Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zekuan Xu, Director of the Department of General Surgery, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JSPH-0504
Record Dates: First submitted 2015-12-30; First posted 2015-12-31 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Roux-en-Y anastomosis (Other): Conventional Roux-en-Y Gastrojejunostomy will be used after laparoscopic distal gastrectomy for early gastric cancer.
  Interventions: Procedure: Conventional Roux-en-Y Gastrojejunostomy
- Uncut Roux-en-Y anastomosis (Experimental): Uncut Roux-en-Y Gastrojejunostomy will be used after laparoscopic distal gastrectomy for early gastric cancer.
  Interventions: Procedure: Uncut Roux-en-Y Gastrojejunostomy

INTERVENTIONS:
Procedure: Conventional Roux-en-Y Gastrojejunostomy — Conventional Roux-en-Y Gastrojejunostomy after laparoscopic distal gastrectomy for early gastric cancer patients
  Arms: Conventional Roux-en-Y anastomosis
Procedure: Uncut Roux-en-Y Gastrojejunostomy — Uncut Roux-en-Y Gastrojejunostomy after laparoscopic distal gastrectomy for early gastric cancer patients
  Arms: Uncut Roux-en-Y anastomosis

SUMMARY:
The current commonly used for distal gastri cancer in gastrointestinal anastomosis is Roux-en-Y. However, the complications after Roux-en-Y reach an incidence of over 30% which involve nausea, vomiting, and abdominal distension. The underlying mechanism might be the result of interruption of intestine peristalsis. In 2013, Kim reported total laparoscopic uncut Roux-en-Y anastomosis could reduce Roux stasis syndrome incidence by keeping the continuity of jejunum. In September 2014, we carried out this operation in 30 cases in our centre. Our previous results showed that this operation had a low postoperative complication and short hospitalization time, indicating uncut Roux-en-Y anastomosis might be a safe procedure. However, some limitations are noticed. The report from South Korea is a retrospective study and the evaluation of QOL is certain subjective. Here, we aimed to perform the first randomized controlled clinical study on uncut Roux-en-Y anastomosis to improve QOL of patients after laparoscopic distal gastrectomy.

DETAILED DESCRIPTION:
The current commonly used for distal gastri cancer in gastrointestinal anastomosis is Roux-en-Y. However, the complications after Roux-en-Y reach an incidence of over 30% which involve nausea, vomiting, and abdominal distension. The underlying mechanism might be the result of interruption of intestine peristalsis. In 2013, Kim reported total laparoscopic uncut Roux-en-Y anastomosis could reduce Roux stasis syndrome incidence by keeping the continuity of jejunum. In September 2014, we carried out this operation in 30 cases in our centre. Our previous results showed that this operation had a low postoperative complication and short hospitalization time, indicating uncut Roux-en-Y anastomosis might be a safe procedure. However, some limitations are noticed. The report from South Korea is a retrospective study and the evaluation of QOL is certain subjective. Here, we aimed to perform the first randomized controlled clinical study on uncut Roux-en-Y anastomosis to improve QOL of patients after laparoscopic distal gastrectomy. The primary aim is to determine whether uncut Roux-en-Y anastomosis improve the quality of life of patients after laparoscopic distal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopy and biopsy confirmed gastric antrum or angle (from the cardia more than 4cm) of gastric cancer
* tumor stage: I
* There is no experience with chemotherapy, no distant metastasis
* Have their own ability to answer the questionnaire
* There is no mental illness
* Age between 18-70 years old
* Agreed to participate in the experiment and signed informed consent

Exclusion Criteria:

* pregnant or nursing patients
* The combined more serious cardiovascular disease, liver and kidney dysfunction (glutamic-pyruvic transaminase/glutamic oxalacetic transaminase more than three times the upper limit of normal, serum creatinine more than 50% higher than the upper limit of normal), abnormal blood clotting function (mean prothrombin time, activated partial thromboplastin time higher than normal values above the upper limit of 50%), neuropsychiatric disorders
* Patients with active infection
* Have other malignant tumor
* Some reason withdraw subjects, can not enrolled in the study again

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Quality of life | one year

SECONDARY OUTCOMES:
Complications | one year

CONTACTS AND LOCATIONS:
Overall Officials: Zekuan Xu, Professor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be open access.

REFERENCES:
- [Derived] Cai Z, Mu M, Ma Q, Liu C, Jiang Z, Liu B, Ji G, Zhang B. Uncut Roux-en-Y reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2024 Feb 29;2(2):CD015014. doi: 10.1002/14651858.CD015014.pub2. PMID 38421211
- [Derived] Xu H, Yang L, Zhang DC, Li Z, Li QY, Wang LJ, Li FY, Wang WZ, Xia YW, Xu ZK. To cut or not to cut? A prospective randomized controlled trial on short-term outcomes of the uncut Roux-en-Y reconstruction for gastric cancer. Surg Endosc. 2023 Aug;37(8):6172-6184. doi: 10.1007/s00464-023-10067-0. Epub 2023 May 9. PMID 37160808